CLINICAL TRIAL: NCT06499428
Title: "Tasso di Stimolazione Ventricolare Nel Follow-up Dei Pazienti Sottoposti ad Impianto di PM Post TAVI:Fattori Predittivi ed Evoluzione Clinica"
Brief Title: Ventricular Pacing Rate in Follow-up of Patients Treated With Definitive PM Implantation Post TAVI
Acronym: P-P-P-TAVI
Status: Active, not recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: P-P-P-TAVI
Record Dates: First submitted 2024-07-05; First posted 2024-07-12 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-04

CONDITIONS: Aortic Stenosis; Conduction Defect, Cardiac
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiac Conduction System Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — brain natriuretic peptide
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the effective ventricular pacing rate in follow-up of patients who underwent a pacemaker (PM) implantation after transcatheter aortic valve implantation (TAVI).

Secondly the study want investigate possible conduction recovery in follow up of patients and possible predictive factors of different ventricular pacing rates.

DETAILED DESCRIPTION:
Aortic stenosis represents the most common valve defect in developed countries. Percutaneous transcatheter aortic valve implantation (TAVI) is now a first-line therapy for aortic stenosis.

The development of conduction blocks remains one of the most frequent complications of TAVI (3-26%), requiring the implantation of a permanent pacemaker (PM).

The damage caused to the conduction system during TAVI is the consequence of the anchoring of the prosthesis to the membranous septum.

There are several clinical, procedural and anatomical variables that correlate with a higher risk of permanent PM implantation post-TAVI, including age, pre-existence of BBDX, development of BBSX post TAVI, use of self-valves -expanding and implantation depth of the bioprosthesis.

Some anatomical variables, obtained from the CT study, appear to correlate with a greater risk of damage to the conduction system post-TAVI.

Recent studies have proven the importance of an accurate measurement of the length of the membranous septum, to design the depth of the bioprosthesis implant while minimizing the risk of damage to the conduction system.

The damage suffered by the conduction system, following the anchoring of the bioprosthesis, is largely inflammatory, and can, as such, be unpredictable in its evolution, and regress over time.

Recent data from the literature suggest that right ventricular stimulation by PM may, in the long term, worsen the prognosis of patients undergoing TAVI, and be associated with a higher rate of mortality from all causes and hospitalizations for decompensation, particularly when the percentage of PM stimulation is > 40%.

Furthermore, post-TAVI permanent PM implantation correlates with increased intensive care and hospitalization times, as well as healthcare costs.

Literature data regarding the evolution of post-TAVI conduction defects are still relatively lacking, and studies regarding the pacing percentage and its impact in post-TAVR patients are limited, especially in the long term, and based on small populations.

According to a recent meta-analysis, approximately half of the patients are not pacemaker dependent 1 year after implantation, furthermore the presence of pre-existing right bundle branch block and the use of self-expanding valves appear to be associated with a doubled risk of developing pacemaker dependence . .

The possibility and time of recovery of the conduction system post TAVI, and, consequently, the need for ventricular pacing, could also depend on some anatomical variables, including the length of the membranous septum and the presence of sub-valvular calcifications

ELIGIBILITY:
Inclusion Criteria:

* PM implantation following TAVI surgery, during the same hospitalization
* Signature of informed consent
* Over the age of 18.

Exclusion Criteria:

* PM implantation prior to hospitalization for TAVI
* PM implantation during hospitalization different from the hospitalization for TAVI
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Data relating to all patients undergoing PM implantation will be collected in the days of hospitalization following TAVI surgery at our current institute (IRCCS Galeazzi Hospital - Sant'Ambrogio) between September 2022 and the closure of the study.
Sampling Method: Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
ventricular pacing rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michela Tarascio, Principal Investigator — IRCCS Galeazzi Sant'Ambrogio
Locations (1):
- IRCCS Ospedale GAleazzi-Sant'Ambrogio, Milan, Italy